CLINICAL TRIAL: NCT01152281
Title: Study to Test Meta-intervention to Increase Retention in HIV Prevention Counseling
Brief Title: Selective Exposure in HIV Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Duval County Health Department (Unknown)
Responsible Party: Principal Investigator, Dolores Albarracin, PhD, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: selectiveexposure
Record Dates: First submitted 2010-05-28; First posted 2010-06-29 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2010-06

CONDITIONS: HIV Infections
Keywords: retention; attrition; empowering; reactance; motivational; goals; Basic control; Control with stories of people with AIDS; Instrumental; Instrumental and Empowering
MeSH Terms: conditions — HIV Infections; Tooth Wear

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Maximal Control (Active Comparator): Basic awareness messages with stories of people living with AIDS
  Interventions: Behavioral: Maximal Control
- Instrumental (Experimental): Instrumental messages with stories of people living with HIV
  Interventions: Behavioral: Instrumental
- Empowering (Experimental): Empowering messages with stories of people living with HIV
  Interventions: Behavioral: Empowering
- Instrumental and Empowering (Experimental): Instrumental and empowering messages with stories of people living with HIV
  Interventions: Behavioral: Instrumental and Empowering
- Minimal Control (Active Comparator): Basic awareness messages with stories of people who are not infected with HIV
  Interventions: Behavioral: Minimal Control

INTERVENTIONS:
Behavioral: Maximal Control — 30 min video with stories of people with HIV. Content describes general health and emotional benefits of counseling.
  Arms: Maximal Control
Behavioral: Instrumental and Empowering — Mix of Instrumental and empowering messages with stories of people living with HIV
  Arms: Instrumental and Empowering
Behavioral: Minimal Control — Control messages to increase awareness of HIV risk
  Arms: Minimal Control
Behavioral: Instrumental — Instrumental messages with stories of people living with HIV
  Arms: Instrumental
Behavioral: Empowering — Empowering messages with stories of people living with HIV
  Arms: Empowering

SUMMARY:
Unfortunately, people most at risk for HIV are the least likely to enroll and remain in prevention programs. In our past work, we have learned how to increase enrollment in such programs among this group. We have identified and addressed previously ignored gender-specific and client self-validation issues that conventional interventions often leave not only uncontrolled, but often biased against participation. The present work will extend these methods from enrollment to retention.

We intend to recruit a sample of 656 at-risk participants through our collaboration with the Duval County, FL Health Department for our randomized, double-blind trial. Our study will investigate if a meta-intervention video designed for empowering participants as agents of their own change can increase the number of attended sessions relative to a control condition without such a video. This trial will also determine if a meta-intervention video addressing various emotional/social and instrumental benefits of an HIV-prevention-counseling intervention can also increase the number of attended sessions. These two factors will be crossed, and their effects on retention will be estimated for different genders and ethnicities. Effects on clients' attention to the return sessions as reported by the counselor will also be explored among participants who return.

We will also conduct mediator analyses for investigating if the meta-intervention has mediating influences on corresponding expectations about the return counseling session. As the inclusion of meta-cognitive measures can alter the efficacy of the intervention, half of the sample will receive measures immediately (0-10 minutes) after exposure to the meta-intervention, before attendance to the next session is registered. The other half will not complete these measures.

DETAILED DESCRIPTION:
1. After the Informed Consent is signed, the research assistant supervises administration of the baseline questionnaire via ACASI. In ACASI, the questions are seen on the computer screen and heard through earphones simultaneously. This technique has been shown to enhance the accuracy of any reported non-normative behavior by the relative privacy and anonymity it affords. It is expected to take about 30 minutes.
2. Participants are seen for one-on-one HIV counseling for approximately 20 minutes by counselors briefed to the study according to the protocol described in the attached document "Scripts Florida Study.doc" (hereinafter "the Scripts document").
3. After the counseling session, participants will watch a 20-minute video delivering one of the experimental or control meta-intervention messages, which are more fully described in the Scripts document.
4. The self-reporting of expectations and intentions that we need to elicit at this point may have a confounding effect on the retention that the study hopes to measure. Therefore, half of the participants will skip the next step and half will complete it, to allow us to assess the actual effect of this self-report measure on retention while studying if these measures mediate retention.
5. The half of the participants reporting expectations will report their expectations and intentions for further counseling, via a 10-minute ACASI questionnaire. The questionnaire is designed to distinguish the dimensions of social/emotional, instrumental and empowering expectations.
6. At the end of the first 70-80 minute session, the counselor schedules the follow-up appointments.
7. Customary phone reminders are issued two days before each 20-minute follow-up session, as is routine for medical and counseling appointments.
8. The study counselor does the following at each follow-up session:

   * Records the participant's attendance or absence on the Counselor's Questionnaire.
   * For attending participants, the study counselor rates their attention to the counseling on the Counselor's Questionnaire.
   * The RA in charge of video presentation rates attention to the videos.
   * At the end of the second session, the study counselor double-checks the third appointment with the participant, and reschedules if necessary.
9. A detailed description of the two follow-up sessions is found in the attached document titled "Counselor Guidelines (2nd and 3rd sessions). The questions and statements therein will be delivered and answered verbally.
10. At the end of the third session, participants who did not answer the questionnaire in Step 5 will answer a similar questionnaire about their reactions to the meta-intervention video.
11. All participants will be fully debriefed. Non-attendees will be called and debriefed either by phone or in person based on their preferences.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active,
* Low condom use,
* Low intention to use condom

Exclusion Criteria:

* Trying to get pregnant
* HIV positive
* with contaminant knowledge about the study
* planning to leave the area

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 722 (Actual)
Dates: Start 2010-05; Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Enrollment | 1 month
  return rate for 2 upcoming sessions

SECONDARY OUTCOMES:
Perceptions of the counselor | 0-10 minutes
  Questionnaire measures of perceptions of the counseling session

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Albarracin, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Duval County Health Department, Jacksonville, Florida, United States

REFERENCES:
- [Background] Albarracin D, Wilson K, Durantini MR, Sunderrajan A, Livingood W. A meta-intervention to increase completion of an HIV-prevention intervention: Results from a randomized controlled trial in the state of Florida. J Consult Clin Psychol. 2016 Dec;84(12):1052-1065. doi: 10.1037/ccp0000139. Epub 2016 Oct 27. PMID 27786499